CLINICAL TRIAL: NCT02402881
Title: Patient-Centered Education Bundle to Decrease Patient Refusal of Venous Thromboembolism (VTE) Prophylaxis
Brief Title: Education Bundle to Decrease Patient Refusal of VTE Prophylaxis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00057117
Record Dates: First submitted 2015-03-25; First posted 2015-03-30 (Estimated); Results first posted 2020-01-06 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2019-12

CONDITIONS: Venous Thromboembolism; Deep Venous Thrombosis; Pulmonary Embolism
Keywords: venous thromboembolism; deep venous thrombosis; pulmonary embolism; blood clots
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism; Thrombosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): A patient-centered education bundle that will be delivered as an in-person, 1-on-1 discussion session with a nurse educator. Supporting education materials include a 2-page patient education sheet and a patient education video.
  Interventions: Behavioral: Patient-centered education bundle
- Control (No Intervention): Patients will receive only the standard practices of care

INTERVENTIONS:
Behavioral: Patient-centered education bundle — A patient-centered education bundle that will be delivered as an in-person, 1-on-1 discussion session with a nurse educator. Supporting education materials include a 2-page patient education sheet and a patient education video.
  Arms: Intervention

SUMMARY:
The investigators have recently developed a registry of missed doses of VTE prophylaxis that includes retrospective data on missed doses of VTE prophylaxis. To decrease rates of VTE prophylaxis refusal, the group has developed a patient-centered education bundle that will be delivered as an in-person, 1-on-1 discussion session with a nurse educator. Supporting education materials include a 2-page education sheet and an educational video.

The investigators hypothesize that patient refusal of VTE prophylaxis is associated with significant knowledge gaps among patients regarding patients' risk of developing VTE and the benefits of VTE prophylaxis and that delivering an education bundle to patients that refuse VTE prophylaxis will improve compliance with VTE prophylaxis and decrease rates of VTE.

DETAILED DESCRIPTION:
Background

This research group's published pilot study reported that nearly 12% of prescribed doses of pharmacologic VTE prophylaxis are not administered and almost 60% of missed doses are due to patient or family member refusal. Fanikos et al found that 44% of missed doses of VTE prophylaxis were due to patient refusal. In a survey of 500 recently hospitalized patients, the National Blood Clot Alliance found that only 28% and 15% respectively had basic knowledge of deep venous thrombosis (DVT) or pulmonary embolism (PE) despite the fact that 15% of participants had a history and 43% had a family history of either condition.

Given these high rates of patient refusal of VTE prophylaxis and significant knowledge gaps regarding VTE, there is an urgent need to educate patients and families on the importance and benefits of compliance with VTE prophylaxis.

The proposed patient-centered education bundle will be delivered as an in-person, 1-on-1 discussion session with a nurse educator. Supporting education materials include a 2-page education sheet and an educational video.

The investigators hypothesize that patient refusal of VTE prophylaxis is associated with significant knowledge gaps among patients regarding patients' risk of developing VTE and the benefits of VTE prophylaxis and that delivering an education bundle to patients that refuse VTE prophylaxis will improve compliance with VTE prophylaxis and decrease rates of VTE.

Objectives

Primary objective: is to determine the impact of delivering a patient education intervention bundle on rates of VTE prophylaxis non-administration.

Secondary objective: is to determine the impact of delivering a patient education intervention bundle on rates of VTE.

Methods

The investigators have developed a real-time alert that notifies a member of the research team whenever a patient misses patients' dose of VTE prophylaxis. This interventional study will take place on on four hospital floors. Whenever a nurse educator receives an alert from any of the included floors indicating that a dose of VTE prophylaxis has been missed, she/he will visit the floor, and approach the nurse in charge of that patient to find out the reason for the missed dose. If the dose was missed as a result of patient refusal, the nurse educator will visit the patient and deliver the education bundle comprised of: 1) a one-on-one education session, 2) the patient education sheet and 3) the patient education video depending on patient preference. The intervention will be in real time for doses missed on business days between 8.00am and 4.00pm and at the start of the next business day for doses missed during non-business hours or on weekends. The investigators anticipate that the study will continue for 5 years and the investigators anticipate a total of 1000 patients during the study duration.

ELIGIBILITY:
Inclusion Criteria:

* All patients on the four trial floors who miss at least one dose of VTE prophylaxis will be included in the study.

Exclusion Criteria:

* N/A

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19652 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliott R Haut, MD PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Medical Institutions, Baltimore, Maryland, United States

REFERENCES:
- [Background] Shermock KM, Lau BD, Haut ER, Hobson DB, Ganetsky VS, Kraus PS, Efird LE, Lehmann CU, Pinto BL, Ross PA, Streiff MB. Patterns of non-administration of ordered doses of venous thromboembolism prophylaxis: implications for novel intervention strategies. PLoS One. 2013 Jun 14;8(6):e66311. doi: 10.1371/journal.pone.0066311. Print 2013. PMID 23799091
- [Background] Fanikos J, Stevens LA, Labreche M, Piazza G, Catapane E, Novack L, Goldhaber SZ. Adherence to pharmacological thromboprophylaxis orders in hospitalized patients. Am J Med. 2010 Jun;123(6):536-41. doi: 10.1016/j.amjmed.2009.11.017. PMID 20569760
- [Background] Maynard GA, Varga EA, Friedman RJ, Brownstein AP, Ansell JE. Deep vein thrombosis and pulmonary embolism: Awareness and prophylaxis practices reported by recently hospitalized patients. Society of Hospital Medicine Annual Meeting. 2011
- [Derived] Owodunni OP, Lau BD, Wang J, Shaffer DL, Kraus PS, Holzmueller CG, Aboagye JK, Hobson DB, Varasteh Kia M, Armocida S, Streiff MB, Haut ER. Effectiveness of a Patient Education Bundle on Venous Thromboembolism Prophylaxis Administration by Sex. J Surg Res. 2022 Dec;280:151-162. doi: 10.1016/j.jss.2022.07.015. Epub 2022 Aug 12. PMID 35969933
- [Derived] Haut ER, Aboagye JK, Shaffer DL, Wang J, Hobson DB, Yenokyan G, Sugar EA, Kraus PS, Farrow NE, Canner JK, Owodunni OP, Florecki KL, Webster KLW, Holzmueller CG, Pronovost PJ, Streiff MB, Lau BD. Effect of Real-time Patient-Centered Education Bundle on Administration of Venous Thromboembolism Prevention in Hospitalized Patients. JAMA Netw Open. 2018 Nov 2;1(7):e184741. doi: 10.1001/jamanetworkopen.2018.4741. PMID 30646370
- See also: PCORI Website Page - "Improving Patient-Nurse Communication to Prevent a Life-Threatening Complication" — http://www.pcori.org/research-in-action/improving-patient-nurse-communication-prevent-life-threatening-complication
- See also: PCORI Website Page - "Preventing Venous Thromboembolism: Empowering Patients and Enabling Patient-Centered Care via Health Information Technology" — http://www.pcori.org/research-results/2013/preventing-venous-thromboembolism-empowering-patients-and-enabling-patient

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 16 medical and surgical hospital units were included, intensive care units were excluded. Convenience sample of 4 units (2 surgical and 2 medical) received the intervention. The remaining 12 units (5 surgical and 7 medical) served as control and received no intervention. Pre-Intervention data were retrospectively assessed
Period: Pre-Intervention Study Period
Arm/Group | Intervention | Control
Started | 2222 | 5657
Completed | 2222 | 5657
Not Completed | 0 | 0
Period: Post-Intervention Study Period
Arm/Group | Intervention | Control
Started | 3111 | 8662
Completed | 3111 | 8662
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention: Patient Visits received the Patient-centered education bundle: A patient-centered education bundle that will be delivered as an in-person, 1-on-1 discussion session with a nurse educator. Supporting education materials include a 2-page patient education sheet and a patient education video.
  This trial treats each visit as a separate enrollment and as a result it is only appropriate to consider the participant at the visit level. The outcomes assessed for this trial were analyzed on the patient visit level, as each visit represents a totally unique participant outcome. For example, Patient A might receive all doses during the first admission to the hospital but the same Patient A might miss doses during a second hospitalization. Similarly, Patient A might have been in Arm 1 during the first hospitalization and in Arm 2 during the second hospitalization.
- Control: Patient Visits received the only the standard practices of care. This trial treats each visit as a separate enrollment and as a result it is only appropriate to consider the participant at the visit level. The outcomes assessed for this trial were analyzed on the patient visit level, as each visit represents a totally unique participant outcome. For example, Patient A might receive all doses during the first admission to the hospital but the same Patient A might miss doses during a second hospitalization. Similarly, Patient A might have been in Arm 1 during the first hospitalization and in Arm 2 during the second hospitalization.
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 5333 | 14319 | 19652
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Each row represents a different period of the study (pre intervention and post intervention) with different number of participants. Overall number of participants represents the number of unique patients in the study. These numbers reflect patient visits at baseline and following the implementation of the patient education intervention.
  Years
    Pre-Intervention: number analyzed (Participants) | 2222 | 5657 | 7879
    Pre-Intervention | 53.9 (17.4) | 56.3 (16.9) | 55.6 (17.1)
    Post-Intervention: number analyzed (Participants) | 3111 | 8662 | 11773
    Post-Intervention | 54.6 (17.6) | 55.8 (16.9) | 55.5 (17.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Each row represents a different period of the study (pre intervention and post intervention) with different number of participants. Overall number of participants represents the number of unique patients in the study. These numbers reflect patient visits at baseline and following the implementation of the patient education intervention.
  Participants
    Pre-Intervention: number analyzed (Participants) | 2222 | 5657 | 7879
    Pre-Intervention: Female | 1153 | 2687 | 3840
    Pre-Intervention: Male | 1069 | 2970 | 4039
    Post-Intervention: number analyzed (Participants) | 3111 | 8662 | 11773
    Post-Intervention: Female | 1587 | 4074 | 5661
    Post-Intervention: Male | 1524 | 4588 | 6112
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Each row represents a different period of the study (pre intervention and post intervention) with different number of participants. Overall number of participants represents the number of unique patients in the study. These numbers reflect patient visits at baseline and following the implementation of the patient education intervention.
  Participants
    Pre-Intervention: number analyzed (Participants) | 2222 | 5657 | 7879
    Pre-Intervention: Black | 941 | 2307 | 3248
    Pre-Intervention: White | 1088 | 2850 | 3938
    Pre-Intervention: Asian | 44 | 117 | 161
    Pre-Intervention: Native American | 9 | 12 | 21
    Pre-Intervention: Others | 140 | 371 | 511
    Post-Intervention: number analyzed (Participants) | 3111 | 8662 | 11773
    Post-Intervention: Black | 1308 | 3469 | 4777
    Post-Intervention: White | 1533 | 4432 | 5965
    Post-Intervention: Asian | 73 | 167 | 240
    Post-Intervention: Native American | 4 | 14 | 18
    Post-Intervention: Others | 193 | 580 | 773
Hospital Unit Type [Count of Participants; unit: Participants] — This refers to the unit of hospital where participants were seen; either surgical or medical units. Population: Each row represents a different period of the study (pre intervention and post intervention) with different number of participants. Overall number of participants represents the number of unique patients in the study. These numbers reflect patient visits at baseline and following the implementation of the patient education intervention.
  Participants
    Pre-Intervention: number analyzed (Participants) | 2222 | 5657 | 7879
    Pre-Intervention: Surgical | 1155 | 2530 | 3685
    Pre-Intervention: Medical | 1067 | 3127 | 4194
    Post-Intervention: number analyzed (Participants) | 3111 | 8662 | 11773
    Post-Intervention: Surgical | 1647 | 4076 | 5723
    Post-Intervention: Medical | 1464 | 4586 | 6050

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Non Administration of Prescribed VTE Prophylaxis Medication Doses
Description: This is the percentage of venous thromboembolism (VTE) prophylaxis doses that were not administered for any reason as documented in the electronic health record by a nurse.
Time Frame: 15 Months
Population: Each row represents a different period of the study (pre intervention and post intervention) with different number of participants. Overall number of participants represents the number of unique patients in the study. These numbers reflect patient visits at baseline and following the implementation of the patient education intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of nonadministration
Arm/Group | Intervention | Control
Number analyzed (Participants) | 5333 | 14319
Percentage of nonadministration
  Pre-Intervention: number analyzed (Participants) | 2222 | 5657
  Pre-Intervention | 9.1 [5.2 to 16.2] | 13.6 [9.8 to 18.7]
  Post-Intervention: number analyzed (Participants) | 3111 | 8662
  Post-Intervention | 5.6 [3.1 to 9.9] | 13.3 [9.6 to 18.5]
Statistical Analysis 1: Comparison: Intervention vs Control; Our primary outcome was the proportion of non-administered doses of prescribed pharmacologic VTE prophylaxis. We compared rates of VTE prophylaxis non-administration pre-post-intervention. For estimating conditional odds ratios (ORs) and their 95% confidence intervals (CIs), the binomial family and a logit link were used; for estimating the conditional proportions, the Poisson family and a log link were used; Test type: Other; p < 0.05, Mixed Models Analysis; We used generalized linear mixed-effects models with multiple outputation reiterated 1000 times to bootstrap the 95% CIs and the P values; Odds Ratio (OR) = 1

2. Secondary Outcome: Number of Participants With Venous Thromboembolism
Description: This is the number of participants with VTE events as documented in the electronic health record.
Time Frame: 15 Months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 5333 | 14319
Participants
  Pre-Intervention: number analyzed (Participants) | 2222 | 5657
  Pre-Intervention | 7 | 14
  Post-Intervention: number analyzed (Participants) | 3111 | 8662
  Post-Intervention | 6 | 17
Statistical Analysis 1: Comparison: Intervention vs Control; Our secondary outcome was the proportion of VTE events. We compared rates of VTE prophylaxis nonadministration pre-post-intervention. For estimating conditional odds ratios (ORs) and their 95% CIs, the binomial family and a logit link were used; for estimating the conditional proportions, the Poisson family and a log link were used; Test type: Other; p < 0.05, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1

ADVERSE EVENTS:
Time Frame: 15 Months
Groups:
- Intervention: Patient Visits received the Patient-centered education bundle: A patient-centered education bundle that will be delivered as an in-person, 1-on-1 discussion session with a nurse educator. Supporting education materials include a 2-page patient education sheet and a patient education video.
- Control: Patient Visits received only the standard practices of care.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/5333 | 0/14319
Serious Adverse Events (participants affected / at risk) | 0/5333 | 0/14319
Other Adverse Events (participants affected / at risk) | 0/5333 | 0/14319

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT02402881/Prot_SAP_000.pdf